CLINICAL TRIAL: NCT05606913
Title: Efficacy and Safety of IBI362 Versus Dulaglutide as add-on to Metformin and/or SGLT2 Inhibitor or TZD in Subjects With Type 2 Diabetes (DREAMS-2)
Brief Title: A Study of IBI362 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI362A302
Record Dates: First submitted 2022-10-19; First posted 2022-11-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBI362 6.0mg (Experimental): ①2mg, SC, once a week* 4weeks; ②4mg, SC, once a week* 4weeks；③6mg, SC, once a week* 20weeks.
  Interventions: Drug: IBI362
- dulaglutide (Experimental): 1.5mg, SC, once a week* 28weeks
  Interventions: Drug: dulaglutide
- IBI362 4.0mg (Experimental): 2mg, SC, once a week* 4weeks; ②4mg, SC, once a week* 24weeks.
  Interventions: Drug: IBI362

INTERVENTIONS:
Drug: dulaglutide — Dulaglutide administered subcutaneously (SC) once a week.
  Arms: dulaglutide
Drug: IBI362 — IBI362 administered subcutaneously (SC) once a week.
  Arms: IBI362 4.0mg; IBI362 6.0mg

SUMMARY:
This trial is conducted in China. The aim of the trial is to evaluate efficacy and Safety of IBI362 Versus dulaglutide as add-on to Metformin and/or SGLT2 inhibitor or TZD in Subjects With Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. T2D was diagnosed according to WHO standards in 1999 for
2. Age ≥ 18 when signing the informed consent form
3. After used stable-dose metformin (≥1500 mg/day) or stable-dose metformin (≥1500 mg/day) combined with SGLT2 inhibitors (empagliflozin 10 mg/day, dapagliflozin 10 mg/day, canagliflozin 100 mg/day, Henagliflozin 5 mg/day) for 2 months before screening, or stable-dose metformin (≥1500 mg/day) combined with daily fixed-dose sulfonylureas (half the maximum dose on the drug label), the blood sugar was still poorly controlled, the local laboratory test at the time of screening was 7.5%≤HbA1c≤11.0%.
4. BMI≥23 kg/m2 at screening.
5. Subjects voluntarily signed the informed consent form and agreed to strictly follow the requirements of this protocol

Exclusion Criteria:

1. Subjects who the investigator thinks may be allergic to the components in the study drug or similar drugs
2. Weight change>5% within 12 weeks before screening (chief complaint)
3. Oral hypoglycemic drugs other than background therapy drugs have been used within 2 months before screening.
4. Previous diagnosis of type 1 diabetes (including adult latent autoimmune diabetes), special type diabetes or gestational diabetes
5. There are active or untreated malignant tumors within 5 years before screening, or patients are in remission of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery)
6. Mental illness existed in the past or at the time of screening, and the researcher thinks it is not suitable to participate in this study
7. Pregnant or lactating women, or men or women who are fertile and unwilling to use contraception throughout the study period
8. The investigator believes that the subject has any other factors that may affect the efficacy or safety evaluation of this study and is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline at week 28 | Baseline, 28 weeks

SECONDARY OUTCOMES:
percent change from baseline in body weigh | Baseline, 28 weeks
Proportion of subjects with HbA1c <7.0% and weight loss ≥5% from baseline | Baseline, 28 weeks
Change from baseline in HbA1c (superiority) | Baseline, 28 weeks
Proportion of subjects with HbA1c <7.0% | Baseline, 28 weeks
Safety,Incidence and severity of adverse events and correlation with study drug; | Baseline to 32weeks
Time to peak plasma concentration (Tmax) | Baseline to 28weeks
Time to peak plasma concentration (Cmax) | Baseline to 28weeks
area under curve (AUC) | Baseline to 28weeks
volume distribution (V) | Baseline to 28weeks
half-life (half-life, T1/2 | Baseline to 28weeks
clearance rate (clearance, CL) | Baseline to 28weeks
To assess changes in PD parameters fasting insulin at different time points before and after administration. | Baseline to 28weeks
To assess changes in PD parameters fasting C-peptide at different time points before and after administration. | Baseline to 28weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijin, China